CLINICAL TRIAL: NCT03571243
Title: Investigation of Oxygenation and Blood Flow in the Brain of Smokers and Their Relation to Smoking Abstinence.
Brief Title: Investigation of Brain Oxygenation and Blood Flow in Smokers
Acronym: OEF
Status: Completed | Type: Observational
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: 44
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Cerebral Oxygenation and Blood Flow in Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smokers: no intervention
  Interventions: Other: no intervention
- never-smokers: no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — observational study

SUMMARY:
Cerebral oxygenation and blood flow in tobacco use disorder and their relation to smoking abstinence will be measured with MRI" ändern in "Cerebral oxygenation and blood flow in tobacco use disorder

DETAILED DESCRIPTION:
In this study, cerebral oxygenation and tobacco-related attentional bias in smokers and non-smokers will be measured with magnetic resonance imaging (MRI).

In this study, the oxygen extraction fraction (OEF), the cerebral blood flow (CBF) and the cerebral metabolic rate of oxygen (CMRO2) are to be measured in smokers and non-smokers using MRI. On the one hand, the influence of chronic smoking (i.e. smokers versus non-smokers) and on the other hand the effect of acute nicotine administration (in smokers) on these parameters will be examined. Furthermore, the influence of these parameters on fMRI results is to be investigated using the example of a stimulus-reaction task. It can be assumed that the OEF does not change through nicotine administration, but differs in smokers and non-smokers and is associated with the strength of tobacco addiction in smokers. CBF and CMRO2 are expected to be reduced in abstinent smokers, but can be normalized by nicotine administration. In this study, 20 smokers and 10 never-smokers will be investigated. Never-smokers will be examined once with MRI and questionnaires, whereas smokers will be examined twice: before and after a smoking break.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* right-handed
* normal or correctable eyesight
* Sufficient ability to communicate with the investigators, to answer questions in oral and written form
* "Fully Informed Consent"
* "Written Informed Consent"
* Group 1 - Smokers: Occasional smoker or tobacco consumption disorder according to DSM 5
* Group 2 - Never-Smokers: Consumption of less than 20 cigarettes in life

Exclusion Criteria:

* women: pregnancy
* Withdrawal of the declaration of consent
* Exclusion criteria for an MRI scan
* severe internal, neurological and psychiatric comorbidities
* Pharmacotherapy with psychoactive substances within the last 14 days
* Current substance abuse
* Axis 1 disorder according to ICD-10 and DSM 5 (except tobacco use disorder and specific phobia within the last 12 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents from Mannheim/Heidelberg Germany and other.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
MRI data | MRI measurement at one day
  oxygenation, blood flow and fMRI data; in smokers pre and post smoking; in never-smokers one session

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Principal Investigator — ZI Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany